CLINICAL TRIAL: NCT05566015
Title: Relationship Between Self-compassion and Treatment Adherence in Schizophrenic Spectrum Disorders
Acronym: CompaSchizo
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Crysalid center Clermont de l'Oise (Unknown); CMP de Montataire (Unknown); CMP de Chambly (Unknown); CMP de Clermont de l'Oise (Unknown); CMP de st Just en Chaussée (Unknown); CMP de Senlis (Unknown); CMP de Crepy en Valois (Unknown); CMP de Pont St Maxence (Unknown); CMP de Chantilly (Unknown); CMP de Creil (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2019_843_0021
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Treatment Adherence; Selfcompassion; Schizophrenic Spectrum Disorder
Keywords: Treatment Adherence; Selfcompassion; schizophrenic spectrum disorder
MeSH Terms: conditions — Treatment Adherence and Compliance | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — self-administered questionnaires as well as clinical assessment of schizophrenia symptoms and depression.

SUMMARY:
Treatment adherence is defined by the World Health Organisation (WHO) as the extent to which the patient's history of therapeutic drug-taking coincides with the prescribed treatment. In patients suffering from psychiatrical diseases, especially in those who are suffering from schizophrenic spectrum disorders, the quality of treatment adherence has to be improved. Indeed, non adherance to anti-psychotic treatment increases the risk of hospitalization, of substance use, violent behaviour and of functionnal and cognitif impairment. Selfcompassion, which involves being touched by and open to one's own suffering and to heal oneself with kindness and without judgement and self-criticism has never beed studied as a possible factor infuencing treatment adherence.

This study aims to evaluate if a link between selfcompassion and treatment adherence exists in patients suffering from schizophrenic spectrum disorders.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with schizophrenia spectrum disorder ( ICD 10 and DSM 5 criteria)
* stabilized (PANNS score under 80)
* aged 18 or above
* In case of tutor or curator, agreement of this person is requiered
* psychiatrist who's following the patient agrees with the study

Exclusion Criteria:

* underage
* non stabilized patient (PANSS score under 80 )
* patient suffering from toxic psychosis
* difficulties to understand french or cognitive impairment which are making it to difficult to answer the different self-administered questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Average level of self compassion | one hour
  The level of self compassion will be assessed with the french version of the Self-compassion scale developped and tested by K.Neff.
  Average scores for the Self-Compassion Scale are around 3.0 on the 1-5 Likert scale, a score of 1-2.5 indicates low self-compassion, 2.5-3.5 indicates moderate, and 3.5-5.0 is an indication of high self-compassion

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No